CLINICAL TRIAL: NCT00206167
Title: A 12-Month Double-Blind, Double-Dummy, Randomized, Parallel Group, Multicenter Efficacy and Safety Study of Symbicort® pMDI 2 x 160/4.5 μg Bid and 2 x 80/4.5 μg Bid Compared to Formoterol Turbuhaler® 2 x 4.5 μg Bid and Placebo in Patients With COPD
Brief Title: A Comparison of Symbicort® pMDI 2 x 160/4.5 μg Bid and 2 x 80/4.5 μg Bid With Formoterol Turbuhaler® 2 x 4.5 μg Bid and Placebo in Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5899C00001; EurodraCT No: 2004-001 168-28; SUN
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide

INTERVENTIONS:
Drug: Budesonide/formoterol pMDI
Drug: Formoterol Turbuhaler

SUMMARY:
The purpose of this study is to compare Symbicort in a pressurized metered-dose inhaler (pMDI) with formoterol and placebo in the long-term maintenance treatment of patients with chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of COPD with symptoms for more than 2 years.
* Smoking history of 10 or more pack years
* A history of at least one COPD exacerbation requiring a course of oral steroids and/or antibiotics within 1-12 months before first visit.

Exclusion Criteria:

* A history of asthma
* Patients taking oral steroids
* Any significant disease or disorder that may jeopardize the safety of the patient

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600
Dates: Start 2005-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Pre-dose and 1-hour post-dose FEV1 over the 12 months treatment period

SECONDARY OUTCOMES:
Patient-reported outcome variables regarding disease status (incl. PEF), collected via questionnaires and diaries
Health care utilization
Safety variables, including adverse events, vital signs, ECG, physical examination, hematology, and clinical chemistry.
all variables assessed over the 12 months treatment period

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Symbicort Medical Science Director, MD, Study Director — AstraZeneca
Locations (216):
- United States (131):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Jasper, Alabama
  - Research Site, Muscle Shoals, Alabama
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Fort Smith, Arkansas
  - Research Site, Carmichael, California
  - Research Site, La Jolla, California
  - Research Site, Lakewood, California
  - Research Site, Los Angeles, California
  - Research Site, Murrieta, California
  - Research Site, Palo Alto, California
  - Research Site, Peninsula, California
  - Research Site, Pismo Beach, California
  - Research Site, Rancho Mirage, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Stockton, California
  - Research Site, Walnut Creek, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, Bay Pines, Florida
  - Research Site, Clearwater, Florida
  - Research Site, DeLand, Florida
  - Research Site, Largo, Florida
  - Research Site, Longwood, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Panama City, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Blue Ridge, Georgia
  - Research Site, Conyers, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Elk Grove Village, Illinois
  - Research Site, Normal, Illinois
  - Research Site, North Chicago, Illinois
  - Research Site, O'Fallon, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Avon, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, Council Bluffs, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, Waterloo, Iowa
  - Research Site, Bowling Green, Kentucky
  - Research Site, Lebanon, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Kenner, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Bangor, Maine
  - Research Site, Taunton, Massachusetts
  - Research Site, Cadillac, Michigan
  - Research Site, Portage, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Missoula, Montana
  - Research Site, McCook, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Scottsbluff, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, Pahrump, Nevada
  - Research Site, Berlin, New Jersey
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Turnersville, New Jersey
  - Research Site, Albany, New York
  - Research Site, Cortland, New York
  - Research Site, Elmira, New York
  - Research Site, Ithaca, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Rochester, New York
  - Research Site, Tonawanda, New York
  - Research Site, High Point, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Chardon, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Mogadore, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Youngstown, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Beaver, Pennsylvania
  - Research Site, Downingtown, Pennsylvania
  - Research Site, Elverson, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Swarthmore, Pennsylvania
  - Research Site, Upland, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Providence, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Union, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Corsicana, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Provo, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Abingdon, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Spokane, Washington
- Bulgaria (5):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Denmark (14):
  - Research Site, Aalborg
  - Research Site, Christiansfeld
  - Research Site, Frederikshavn
  - Research Site, Frederikssund
  - Research Site, Hellerup
  - Research Site, Kobenhavn K
  - Research Site, København N
  - Research Site, København NV
  - Research Site, København S
  - Research Site, Silkeborg
  - Research Site, Skive
  - Research Site, Svendborg
  - Research Site, Viborg
  - Research Site, Værløse
- Germany (26):
  - Research Site, Cottbus, Brandenburg
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Münster, North Rhine-Westphalia
  - Research Site, Dresden, Saxony
  - Research Site, Jena-Maua, Thuringia
  - Research Site, Bad Salzungen
  - Research Site, Bad Segeberg
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Cologne
  - Research Site, Erfurt
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Geesthacht
  - Research Site, Gelnhausen
  - Research Site, Gelsenkirchen
  - Research Site, Grobhansdorf
  - Research Site, Hanover
  - Research Site, Kassel
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Neuruppin
  - Research Site, Potsdam
- Greece (4):
  - Research Site, Athens
  - Research Site, Hraklion- Crete
  - Research Site, Larissa
  - Research Site, Thessaloniki
- Hungary (28):
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Deszk
  - Research Site, Érd
  - Research Site, Füzesabony
  - Research Site, Godolli
  - Research Site, Gyöngyös
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Jászberény
  - Research Site, Keszthely
  - Research Site, Kiskunhalas
  - Research Site, Mosdós
  - Research Site, Mosonmagyaróvár
  - Research Site, Nógrádgárdony
  - Research Site, Pécs
  - Research Site, Salgótarján
  - Research Site, Sárvár
  - Research Site, Siófok
  - Research Site, Szarvas
  - Research Site, Százhalombatta
  - Research Site, Szeged
  - Research Site, Szombathely
  - Research Site, Tatabánya
  - Research Site, Törökbálint
  - Research Site, Veszprém
  - Research Site, Zalaegerszeg
  - Research Site, Zalaegerszeg-Pozva
- Research Site, Reykjavik, Iceland
- Mexico (3):
  - Research Site, Mexico City, D.F.
  - Research Site, Guadalajara, Jalisco
  - Research Site, Monterrey, Nuevo León
- Romania (4):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Deva
  - Research Site, Iași

REFERENCES:
- [Derived] Bafadhel M, Peterson S, De Blas MA, Calverley PM, Rennard SI, Richter K, Fageras M. Predictors of exacerbation risk and response to budesonide in patients with chronic obstructive pulmonary disease: a post-hoc analysis of three randomised trials. Lancet Respir Med. 2018 Feb;6(2):117-126. doi: 10.1016/S2213-2600(18)30006-7. Epub 2018 Jan 10. PMID 29331313
- [Derived] Make BJ, Eriksson G, Calverley PM, Jenkins CR, Postma DS, Peterson S, Ostlund O, Anzueto A. A score to predict short-term risk of COPD exacerbations (SCOPEX). Int J Chron Obstruct Pulmon Dis. 2015 Jan 27;10:201-9. doi: 10.2147/COPD.S69589. eCollection 2015. PMID 25670896
- [Derived] Bleecker ER, Meyers DA, Bailey WC, Sims AM, Bujac SR, Goldman M, Martin UJ. ADRB2 polymorphisms and budesonide/formoterol responses in COPD. Chest. 2012 Aug;142(2):320-328. doi: 10.1378/chest.11-1655. PMID 22383665